CLINICAL TRIAL: NCT01490827
Title: Argus® II Retinal Prosthesis System Post-Market Surveillance Study
Status: Terminated | Type: Observational
Why Stopped: Sponsor discontinued the Argus II product
Sponsor: Second Sight Medical Products (Industry)
Responsible Party: Sponsor
Other Study IDs: PM-01
Record Dates: First submitted 2011-12-05; First posted 2011-12-13 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Outer Retinal Degeneration; Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Argus II Retinal Prosthesis: Patients implanted with an Argus II Retinal Prosthesis

SUMMARY:
This post-market surveillance study is conducted in the European Economic Area where Argus II has been CE certified for use in outer retinal degeneration patients.

DETAILED DESCRIPTION:
This study is being conducted to monitor the use of Argus II in a larger population than available within pre-market approval studies. Safety data will be monitored to ensure continued acceptability of risks to study participants, and an attempt will be made to include all eligible and willing participants implanted with Argus II. Measures of visual function that may contribute to device improvements will also be gathered and evaluated.

ELIGIBILITY:
Inclusion Criteria:

Adults, age 25 year or older

* with severe to profound outer retinal degeneration (not including Age-related Macular Degeneration)
* Have some residual light perception. If no residual light perception remains, the retina must be able to respond to electrical stimulation;
* Have previous history of useful form vision
* Have consented to participate in the study
* Had an Argus II Retinal Prosthesis surgically implanted 14 days (± 7 days) prior to enrollment (at Baseline Visit) in the study
* At the time of the Baseline Visit, do not suffer from non-ophthalmic serious adverse events (e.g. coma, myocardial infarction, etc.).

Exclusion Criteria:

* Ocular diseases or conditions that could prevent Argus II from working (e.g. optic nerve disease, central retinal artery or vein occlusion, history of retinal detachment, trauma, severe strabismus, etc.)
* Ocular structures or conditions that could prevent the successful implantation of the Argus II Implant or adequate healing from surgery (e.g. extremely thin conjunctiva; axial length <20.5 mm or > 26 mm; corneal ulcers; choroidal neovascularization in the area of the intended tack location, etc.)
* Ocular diseases or conditions (other than cataracts) that prevent adequate visualization of the inner structures of the eye (e.g. corneal opacity)
* Pre-disposition to eye rubbing
* Any disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocols, including:

  * cognitive decline including diagnosed forms of dementia and/or progressive neurologic disease,
  * psychiatric disease including diagnosed forms of depression;
  * does not speak a principal language associated with the region, and
  * deafness or selective frequency hearing loss that prevents hearing device alarms and alerts
* Participants who are pregnant or wish to become pregnant during the course of the study
* Participation in another investigational drug or device study that may conflict with the objectives, follow-up or testing of this study;
* Conditions likely to limit life to less than 1 year from the time of inclusion.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from eligible patients who have been implanted with the Argus II retinal prosthesis at the enrolling center.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
adverse events | up to 3 years from time of implantation
  nature and rate of adverse events

SECONDARY OUTCOMES:
visual function | up to 3 years from time of implantation
  Square localization, direction of motion, grating visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Ripley, Study Director — Second Sight Medical Products
Locations (10):
- Germany (8):
  - Augenklinik des Staedtischen Klinikums, Karlsruhe, Baden-Wurttemberg
  - Klinikum rechts der Isar - Technical University, Munich, Bavaria
  - Center for Ophthalmology - University of Koln, Cologne, North Rhine-Westphalia
  - Knappschaftsklinikum Saar, Department of Ophthalmology, Sulzbach, Saarland
  - University Medical Center Schleswig-Holstein, Department of Ophthalmology, Lübeck, Schleswig-Holstein
  - RWTH University Eye Clinic, Aachen
  - University Hospital Hamburg-Eppendorf, Klinik u. Poliklinik fur Augenheilkunde, Hamburg
  - Universitätsklinikum Leipzig AöR, Klinik und Poliklinik für Augenheilkunde, Leipzig
- Italy (2):
  - University of Pisa Eye Surgery Department, Pisa, Tuscany
  - ULSS 15 Alta Padovana Hospital, Camposampiero, Veneto

REFERENCES:
- [Background] da Cruz L, Coley BF, Dorn J, Merlini F, Filley E, Christopher P, Chen FK, Wuyyuru V, Sahel J, Stanga P, Humayun M, Greenberg RJ, Dagnelie G; Argus II Study Group. The Argus II epiretinal prosthesis system allows letter and word reading and long-term function in patients with profound vision loss. Br J Ophthalmol. 2013 May;97(5):632-6. doi: 10.1136/bjophthalmol-2012-301525. Epub 2013 Feb 20. PMID 23426738
- [Background] Weiland JD, Faraji B, Greenberg RJ, Humayun MS, Shellock FG. Assessment of MRI issues for the Argus II retinal prosthesis. Magn Reson Imaging. 2012 Apr;30(3):382-9. doi: 10.1016/j.mri.2011.12.005. Epub 2012 Jan 20. PMID 22260934
- [Result] Schaffrath K, Schellhase H, Walter P, Augustin A, Chizzolini M, Kirchhof B, Grisanti S, Wiedemann P, Szurman P, Richard G, Greenberg RJ, Dorn JD, Parmeggiani F, Rizzo S. One-Year Safety and Performance Assessment of the Argus II Retinal Prosthesis: A Postapproval Study. JAMA Ophthalmol. 2019 Aug 1;137(8):896-902. doi: 10.1001/jamaophthalmol.2019.1476. PMID 31145440
- [Derived] Gregori NZ, Callaway NF, Hoeppner C, Yuan A, Rachitskaya A, Feuer W, Ameri H, Arevalo JF, Augustin AJ, Birch DG, Dagnelie G, Grisanti S, Davis JL, Hahn P, Handa JT, Ho AC, Huang SS, Humayun MS, Iezzi R Jr, Jayasundera KT, Kokame GT, Lam BL, Lim JI, Mandava N, Montezuma SR, Olmos de Koo L, Szurman P, Vajzovic L, Wiedemann P, Weiland J, Yan J, Zacks DN. Retinal Anatomy and Electrode Array Position in Retinitis Pigmentosa Patients After Argus II Implantation: An International Study. Am J Ophthalmol. 2018 Sep;193:87-99. doi: 10.1016/j.ajo.2018.06.012. Epub 2018 Jun 27. PMID 29940167
- [Derived] Rizzo S, Belting C, Cinelli L, Allegrini L. Visual field changes following implantation of the Argus II retinal prosthesis. Graefes Arch Clin Exp Ophthalmol. 2015 Feb;253(2):323-5. doi: 10.1007/s00417-014-2822-0. Epub 2014 Nov 30. No abstract available. PMID 25432093
- [Derived] Olson JL, Velez-Montoya R, Mandava N, Stoldt CR. Intravitreal silicon-based quantum dots as neuroprotective factors in a model of retinal photoreceptor degeneration. Invest Ophthalmol Vis Sci. 2012 Aug 17;53(9):5713-21. doi: 10.1167/iovs.12-9745. PMID 22761263